CLINICAL TRIAL: NCT04170309
Title: Retrospective Chart Review to Evaluate the Safety Profile of Ceftobiprole in Patients With Impaired Hepatic or Renal Function or Immunosuppression
Brief Title: Collection of Data of Ceftobiprole Treated Patients: Comparison of Patients With and Without Certain Diseases
Acronym: RETRACE
Status: Completed | Type: Observational
Sponsor: Advanz Pharma (Industry)
Collaborators: AMS Advanced Medical Services GmbH (Industry); APCER Life Sciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: BPR-PAS-001; EUPAS30444 (Other: EU PAS Register)
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Renal Insufficiency; Hepatic Insufficiency; Immunosuppression
Keywords: Cephalosporins; Retrospective Studies; Safety
MeSH Terms: conditions — Renal Insufficiency; Hepatic Insufficiency | interventions — ceftobiprole medocaril

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With medical condition of interest: Participants treated with ceftobiprole with at least one of the following conditions:
  * Renal Insufficiency
  * Hepatic Insufficiency
  * Immunosuppression
  Interventions: Drug: Ceftobiprole medocaril
- Without medical condition of interest: Patients treated with ceftobiprole without any of the following conditions:
  * Renal Insufficiency
  * Hepatic Insufficiency
  * Immunosuppression
  Interventions: Drug: Ceftobiprole medocaril

INTERVENTIONS:
Drug: Ceftobiprole medocaril — Participants in whom treatment with Ceftobiprole medocaril has been completed

SUMMARY:
In this observational study, data from patients treated with the antibiotic ceftobiprole in the past will be collected. The sponsor of the study is Correvio International Sárl, based in Switzerland. Correvio has committed to the health authorities to obtain further information on possible side effects especially in patients suffering from impaired liver or renal function or immune system deficiency and compare these effects to the ones observed in patients without these health problems. Patient data are collected from historic patient charts, patients will not be treated for the purpose of this data collection. All efforts are being made to capture the data of all patients who meet the inclusion criteria and have received at least one dose of ceftobiprole since this drug was first prescribed at the site.

DETAILED DESCRIPTION:
Rationale and background:

Ceftobiprole is a beta-lactam antibiotic with bactericidal activity against a broad spectrum of Gram-positive and Gram-negative bacteria, that was developed to treat patients with pneumonia both in a hospital or community setting. Clinical trials were conducted in adult immune-competent patients with normal or mild to moderate renal or hepatic function impairment. The clinical trial program completed to date has excluded patients with immune suppression and significant organ function impairment (hepatic or renal). The safety profile of ceftobiprole in these patient groups was recognized during the marketing authorization procedure as important missing information and the applicant committed to conduct a post authorization safety study.

A randomized Phase 3 study in the indication of acute bacterial skin and skin structure infections (ABSSSIs) is completed (NCT03137173), and a randomized Phase 3 study in the indication of S. aureus bacteremia is ongoing (NCT03138733). This retrospective chart review is conducted to further evaluate the safety profile of ceftobiprole in patient populations with specific risk factors.

Research question:

To estimate the proportion and the relative frequency of treatment-emergent adverse events (AEs) and adverse event of special interest will be assessed in patients treated with ceftobiprole and who have at least one of the following conditions:

* Impaired renal function
* Impaired hepatic function
* Immunosuppression

Treatment-emergent AEs are defined as events occurring after first study-drug administration, up to 28 days after the completion of treatment.

Adverse Events of Special Interest are the following;

* Hyponatraemia
* Hepatobiliary disorders
* Renal toxicity (including potential interactions with nephrotoxic drugs)
* Coombs test (DAT) positivity + clinical evidence of haemolysis
* Hypersensitivity reactions, including anaphylactic reactions
* Pseudomembranous colitis / C. difficile colitis
* Convulsions

The observed frequency of adverse events and adverse events of special interest in patients with the above risk factors will be compared to the frequency of these adverse events and adverse events of special interest in patients without these risk factors.

The study will enroll patients in whom treatment with ceftobiprole has been completed.

Patient charts will be selected from hospital sentinel sites.

Patient observation would normally be planned for 28 days after completion of ceftobiprole therapy. If, at the time of the review of any patient medical records, an AE has not been resolved, these patients would be followed up until resolution.

The study would continue until the target number of patients has been reached. The end date of this study would be set at the date of the last patient record review, or in cases where follow-up is extended beyond this period, until the end of follow-up.

Variables:

The following variables will be identified from the patient charts

* Year of birth and gender
* Weight
* Indication of treatment
* Attribution to a specific population group (see inclusion criteria) and criteria to assign the patient
* Start date of ceftobiprole
* Stop date of ceftobiprole and main reason for stopping (if known)
* Prescribed dose/regimen at treatment start
* Changes in dose during treatment
* Relevant medical history (diagnosis within 1 year prior to treatment start)
* Presence of ascites and hepatic encephalopathy at baseline
* Laboratory investigations undertaken as part of routine clinical practice and management of the patient related to the outcomes of interest, e.g., serum sodium, AST (aspartate aminotransferase), ALT (alanine aminotransferase), serum albumin, total bilirubin, GGT (gamma-glutamyltransferase) and AP (alkaline phosphatase), prothrombin time, INR (international normalized ratio), creatinine, haemoglobin, HCT (hematocrit), Coombs (DAT), C. difficile toxin tests prior (within 1 month) and up to 28 days after completion of treatment
* Findings of colonoscopy/sigmoidoscopy (for C. difficile colitis)
* Concomitant medication at baseline and up to 28 days after completion of treatment with focus on new onset use or dose modification of medications to treat hypersensitivity/anaphylaxis, convulsions, or C. difficile colitis
* Treatment-emergent AEs (event reports up to 28 days after completion of treatment), with focus on AEs of special interest (AESIs)
* Date and cause(s) of death (if applicable)
* Use during pregnancy (with follow-up until delivery)

Data sources:

This study will use data from patient charts, which includes physician and nurse notes, admission and discharge summaries, consultancy reports, laboratory test sheets, and microbiology sheets.

ELIGIBILITY:
The study will enroll participants in whom treatment with ceftobiprole has been completed (including both on-label and off-label use) plus at least one of the following criteria (more than one criterion may apply):

* Participants with severe renal impairment / ESRD (end-stage renal disease, defined as calculated CLCr ( creatinine clearance) < 30 mL/minute or oliguria < 20 mL/hour unresponsive to fluid challenge or any form of dialysis)
* Impaired baseline hepatic function (patients with liver failure/cirrhosis Child Pugh Grade A, B, C or existing non-cirrhotic liver disease associated with total bilirubin > 2 mg/dL or alanine aminotransferase [ALT], or aspartate aminotransferase [AST] ≥ 3 times upper limit of the normal range [ULN])
* Participants with immunosuppression, i.e.,

  * HIV-positive with CD4 (cluster of differentiation 4) counts of ≤ 0.2 × 10E9/L (≤ 200 cells/mm3)
  * Immunocompromised as determined by the investigator (any type or aetiology)
  * Baseline neutropenia or baseline myelosuppression, defined as presence of myelosuppression or neutropenia (absolute neutrophil count [ANC] ≤ 0.5 × 10E9/L [< 500 polymorphonuclear neutrophils (PMNs)/mm3]), severe anaemia (haemoglobin < 6.5 g/dL), or severe thrombocytopenia (< 49.9 × 10E9/mm3) In addition, the study will enroll a control group of patients in whom treatment has been completed without any of the criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants from hospitals.
Sampling Method: Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Estimation of the proportion and relative frequency of treatment-emergent AEs and AEs of special interest | during and until 28 days after completion of ceftobiprole therapy
Assessment of hyponatraemia | during and until 28 days after completion of ceftobiprole therapy
Assessment of hepatobiliary disorders | during and until 28 days after completion of ceftobiprole therapy
Assessment of renal toxicity (including potential interactions with nephrotoxic drugs) | during and until 28 days after completion of ceftobiprole therapy
Assessment of Coombs test (DAT) positivity + clinical evidence of haemolysis | during and until 28 days after completion of ceftobiprole therapy
Assessment of hypersensitivity reactions, including anaphylactic reactions | during and until 28 days after completion of ceftobiprole therapy
Assessement of Pseudomembranous colitis / Clostridium difficile colitis | during and until 28 days after completion of ceftobiprole therapy
Assessment of convulsions | during and until 28 days after completion of ceftobiprole therapy

SECONDARY OUTCOMES:
Adverse events by indication | during and until 28 days after completion of ceftobiprole therapy
Treatment dosage | During ceftobiprole therapy
Treatment duration in days | During ceftobiprole therapy

CONTACTS AND LOCATIONS:
Overall Officials: Noëlle Jemmely, Study Director — ADVANZ PHARMA Switzerland Sàrl
Locations (18):
- France (2):
  - Montpellier Hopital Lapeyronie, Montpellier
  - Centre Hospitalier de Valenciennes, Valenciennes
- Lungenklinik Neustadt GmbH, Neustadt/Harz, Germany
- Italy (8):
  - Ospedale Sant'Orsola Malpighi, Bologna
  - AORN Ospedali dei Colli - Ospedale 'V. Monaldi, Napoli
  - Policlinico federico II, Napoli
  - AO di Perugia -Ospedale Santa Maria della Misericordia, Perugia
  - AOU Pisana-Cisanello, Pisa
  - AAS n 5 "Friuli Occidentale - Ospedale Santa Maria degli Angeli, Pordenone
  - AOU Città della Salute e della Scienza Torino - Presidio Molinette, Torino
  - ASST Settelaghi - Ospedale di Circolo e Fondazione Macchi, Varese
- Spain (7):
  - Hospital Clínic de Barcelona, Clinical Research Infectious Disease Department (CRID), Barcelona
  - Hospital Universitari MútuaTerrassa Planta 15, Barcelona
  - Servei de Malalties Infeccioses Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario Virgen de las Nieves, 4ª Planta Izquierda, Granada
  - Hospital Central de la Defensa "Gomez Ulla" Planta 22, Madrid
  - Hospital La Moraleja, Madrid
  - Hospital Universitario y Politécnico La Fe Servicio de Neumología. Torre E piso 4º, Valencia

IPD SHARING:
Plan to Share IPD: No